CLINICAL TRIAL: NCT06174376
Title: A Prospective, Multi-Center, Early Feasibility Study to Assess Clinical Outcomes of the GORE Synthetic Cornea Device in Patients With Loss of Corneal Clarity
Brief Title: Clinical Outcomes of the Gore Synthetic Cornea Device
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: W.L.Gore & Associates (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: GSC 23-01
Record Dates: First submitted 2023-12-08; First posted 2023-12-18 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-12

CONDITIONS: Corneal Opacity
Keywords: Artificial Corneal transplantation, corneal opacity, corneal blindness
MeSH Terms: conditions — Corneal Opacity

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- GORE Synthetic Cornea Device (Experimental): Treatment with GORE Synthetic Cornea Device
  Interventions: Device: GORE Synthetic Cornea Device

INTERVENTIONS:
Device: GORE Synthetic Cornea Device — Treatment with GORE Synthetic Cornea Device

SUMMARY:
Study objective is to evaluate the initial safety and effectiveness of the GORE Synthetic Cornea Device in the treatment of loss of corneal clarity in patients who are candidates for corneal transplantation

DETAILED DESCRIPTION:
This is a prospective, single-arm, open-label, multi-center early feasibility clinical study designed to evaluate the clinical outcomes of the GORE Synthetic Cornea Device in the treatment of loss of corneal clarity in patients who are candidates for corneal transplantation.

Following procedure, clinical follow up will be scheduled over the course of the study duration (12 months).

ELIGIBILITY:
Key Inclusion Criteria:

* Patients must meet all of the following criteria to be eligible to be consented for this study.

  1. Patient must be able to comprehend the study requirements and provide written informed consent. Patients must be willing to follow study instructions, agree to comply with all study procedures , and able to return for all scheduled follow-up examinations for 12 months postoperatively (the study duration). The follow-up exams may be extended up to 60 months post operatively if the patient consents to the extension.
  2. Male or female patients ≥ 18 years old at the time of consent
  3. Physical condition suitable for undergoing surgery, as evidenced by medical history and physical examination provided by a licensed medical provider (primary care physician, nurse practitioner, internal medicine physician etc.)
  4. Currently with an opaque cornea (as determined by the investigator) with or without a prior history of failed donor corneal transplantation [penetrating keratoplasty (PK) or endothelial keratoplasty (EK)] and loss of corneal clarity
  5. Best corrected distance visual acuity of worse than 20/400 in the study eye using Snellen chart
  6. Best corrected distance visual acuity of better than 20/200 in the fellow (non-study) eye using Snellen chart
  7. Pseudophakia status in the study eye with a stable posterior chamber intraocular lens (IOL) implant centered within the capsular bag or sulcus
  8. Corneal thickness measurement in study eye (epithelium to endothelium; central and mid-peripheral/ 3 to 5mm away from center at superior, inferior, nasal and temporal quadrants) with each measurement between 700um - 900um, measured using ultrasound (US) pachymetry. If one or more measurements cannot be obtained using US pachymetry, measurements using anterior segment optical coherence tomography (OCT) may be used (with the measurement being between 700-900um)
  9. If applicable, prior corneal transplant ≥ 8 mm in diameter
  10. Adequate lid function and normal ocular surface and tear film parameters for implant of the study device, as determined by the investigator.

Key Exclusion Criteria:

* Patients who meet any of the following exclusion criteria cannot be consented and included in this study:

  1. Inability to provide written informed consent and comply with study assessments for the full duration of the study.
  2. Age: < 18 years
  3. Patients who are pregnant/nursing or planning to become pregnant during the study.

     Note: For women of child-bearing potential, confirmation of pregnancy status must be documented per site standard.
  4. Corneal thickness measurement (epithelium to endothelium; central and mid-peripheral/ 3 to 5mm away from center at superior, inferior, nasal and temporal quadrants) in the study eye with any measurement less than 700um or more than 900um measured using US pachymetry. If one or more measurements cannot be obtained using US pachymetry, measurements using anterior segment OCT may be used
  5. If applicable, prior corneal transplant < 8 mm in diameter
  6. Aphakic or phakic status of the study eye
  7. Pseudophakic status of the study eye with anterior chamber IOL or unstable posterior chamber IOL, according to clinical history or UBM
  8. Evidence of tear film, ocular surface or lid abnormalities in the study eye

     * Schirmer test without anesthesia less than 5 mm at 5 minutes. NOTE: Patient can be eligible after successful tear duct blockage (such as plugs or cauterization) if the Schirmer's are adequate following the procedure
     * Evidence of conjunctival or lid margin keratinization
     * Presence of cicatrizing conjunctivitis (Stevens Johnson Syndrome, mucous membrane pemphigoid, trachoma, chemical, radiation or thermal trauma
     * Prior history of stage II or III neurotrophic keratitis / keratopathy
     * Limbal stem cell deficiency leading to prior episode(s) of recurrent or persistent corneal epithelial defects
     * Prior history of immune-mediated/ non-infectious keratolysis with or without underlying systemic disease
     * Significant lid margin disease with infestation/infection within 30 days prior to surgery.

     NOTE: Patient can be eligible after successful treatment and resolution
     * Significant anatomical lid problems (trichiasis, entropion, ectropion, lagophthalmos, exophthalmos, Bell's palsy, or significant ptosis)
  9. Current or history of corneal or ocular surface infection in the study eye within 30 days prior to surgery.

     NOTE: Patient can be eligible after successful treatment and resolution as determined by the investigator
  10. Any known intolerance or hypersensitivity to topical anesthetics, mydriatics, post-operative antibiotic or steroid drops , topical intraocular pressure lowering drops, allergy to sulfa drugs, or inability to tolerate oral intraocular pressure lowering drugs, or any component of the device
  11. History of ocular or periocular malignancy in the study eye within the previous five years
  12. Current or prior history of herpes simplex virus (HSV) or Varicella-zoster virus (VZV) keratitis in the study eye.
  13. History of shingles vaccination in the past year or intent to receive the vaccine during the study period
  14. Current or prior history of uveitis in the study eye
  15. Current or prior history of scleritis or retinitis in the study eye
  16. Uncontrolled glaucoma defined by having one or both of the below:

      * Intraocular pressure of greater than 21 mm Hg
      * Intraocular pressure above the specific target pressure for the patient NOTE: Patients with history of glaucoma who are on topical glaucoma medications or who have undergone glaucoma surgery with intraocular pressure within the target range are eligible
  17. Hypotony in the study eye, as evidenced by an intraocular pressure of < 6 mmHg
  18. Presence of broad anterior synechia greater than a quadrant, defined by having both of the below:

      * 3 contiguous clock hours of synechia
      * Involving the central 8 mm of the cornea
  19. Presence of significant corneal stromal vascularization, defined by having both of the below:

      * 3 contiguous clock hours of vascularization
      * Involving the central 8 mm of the cornea
  20. Retinal detachment within 30 days prior to surgery. NOTE: Patients with a prior history of retinal detachment surgery are eligible, unless they currently have silicone oil in the posterior segment
  21. Current (or prior) history of other keratoprosthesis device implantation
  22. Monocular status
  23. Inability to wear a soft contact lens due to conjunctival or lid abnormalities
  24. Signs of current (within the two weeks prior to surgery) systemic infection, including fever and current treatment with antibiotics
  25. Participation in another simultaneous interventional medical investigation or trial that may have a reasonable likelihood of affecting the outcomes of the present study
  26. Have any other history of clinically severe diseases, or conditions that in the opinion of the investigator, may affect the results of the study
  27. Any current or history of substance abuse, psychiatric disorder or a condition that, in the opinion of the investigator, may invalidate communication or adherence to study procedures
  28. Patients who are unable to comply with the study procedures and follow-up visits throughout the study period (12 months)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-08-19 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Primary Effectiveness: Device retention | Through 12 months
  Number of study eyes with GORE Synthetic Cornea Device present
Primary Safety: Intraoperative Adverse Events | At Initial Procedure
  Number of subjects with procedure- and/or device-related adverse event during implant procedure
Primary Safety: Post-operative ophthalmic Adverse Events | Through 12 months
  Number of subjects with post-operative ophthalmic adverse event in the study eye
Primary Safety: Secondary surgical Intervention | Through 12 months
  Number of subjects requiring post-operative secondary surgical interventions (SSIs)

SECONDARY OUTCOMES:
Secondary Effectiveness: Improvement in Visual Acuity | Through 12 month
  Number of study eyes with improvement of two lines or more in Best Spectacle Corrected Distance Visual Actuity compared to pre-operative baseline

CONTACTS AND LOCATIONS:
Overall Officials: Arturo Ramirez Miranda, MD, Principal Investigator — Instituto de Oftalmología Fundación de Asistencia Privada Conde Valenciana I.A. P.; Valeria Sanchez Huerta, MD, Principal Investigator — Asociación para Evitar la Ceguera en México, I.A.P
Locations (2):
- Mexico (2):
  - Asociación para Evitar la Ceguera en México, I.A.P, Mexico City
  - Instituto de Oftalmología Fundación de Asistencia Privada Conde Valenciana I.A. P., Mexico City

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ramirez-Miranda A, Ortiz-Morales G, Domene-Hickman JL, Fabregas-Sanchez-Woodworth D, Garcia-Padilla L, Navas A, Akpek EK, Graue-Hernandez EO. Surgical Considerations for the Human Implantation of the Gore Synthetic Corneal Device. Cornea. 2025 Nov 1;44(11):1426-1430. doi: 10.1097/ICO.0000000000003950. Epub 2025 Aug 14. PMID 40810416